CLINICAL TRIAL: NCT03131297
Title: Multicenter Prospective Evaluation of Radiofrequency for Anal Fistulas
Acronym: RADIOFIST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: F Care Systems NV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 17LAZ_RadioFist
Record Dates: First submitted 2017-04-06; First posted 2017-04-27 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Anal Fistula
Keywords: anal fistulas; evaluation of radiofrequency
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anal fistula treated by radiofrequency (Experimental): treatment by radiofrequency: patient with anal fistula treated by radiofrequency
  Interventions: Procedure: treatment by radiofrequency

INTERVENTIONS:
Procedure: treatment by radiofrequency — Radiofrequency might destroy fistula tract without lesion of anal sphincter.

SUMMARY:
Anal fistula treatment is associated with increasing risk of anal incontinence until 40% of cases. New and alternative treatments (glue, advancement flap, plug…) decrease this risk, but with fistula efficacy treatment in 40 to 60% of cases. Radiofrequency might destroy fistula tract without lesion of anal sphincter.

Objective : Fistula healing rate and anal continence, 6 and 12 months after radiofrequency procedure.

Methods : Clinical and MRI evaluation before, 6 and 12 months after treatment. Patients : 50 patients with low, high, complex and Crohn disease fistula. An intermediate analysis is expected after the first 20 patients, to verify morbidity.

Evaluations :

* Fistula clinical healing 6 and 12 months after procedure
* Fistula MRI healing 12 months after procedure
* Anal continence before and after procedure
* Feasibility og radiofrequency procedure
* Morbidity
* Success and failure prognostics factors of this procedure

DETAILED DESCRIPTION:
: Anal fistula treatment is associated with increasing risk of anal incontinence until 40% of cases. New and alternative treatments (glue, advancement flap, plug…) decrease this risk, but with fistula efficacy treatment in 40 to 60% of cases. Radiofrequency might destroy fistula tract without lesion of anal sphincter.

Objective : Fistula healing rate and anal continence, 6 and 12 months after radiofrequency procedure.

Methods : Clinical and MRI evaluation before, 6 and 12 months after treatment. Patients : 50 patients with low, high, complex and Crohn disease fistula. An intermediate analysis is expected after the first 20 patients, to verify morbidity.

Evaluations :

* Fistula clinical healing 6 and 12 months after procedure
* Fistula MRI healing 12 months after procedure
* Anal continence before and after procedure
* Feasibility og radiofrequency procedure
* Morbidity
* Success and failure prognostics factors of this procedure

Schedule :

* First inclusion march 2017
* Last inclusion march 2018
* Evaluations until march 2019.

ELIGIBILITY:
Inclusion Criteria:

* Adult Patient agreeing to participate in the study and signing the consent to participate
* Patients with an anal fistula previously drained, without diverticulum> 10 mm in MRI after drainage.
* For women of childbearing age, they must have a negative urine pregnancy test

Exclusion Criteria:

* Patient minor,
* Patients who are linguistically or psychologically unable to understand the information given and to give informed consent,
* Patient incapable, in the opinion of the investigator, to complete the self-questionnaires,
* Against-indication to radiofrequency treatment (infectious anal pathologies, anal fissures, residual staples of previous treatment Longo,
* Pregnant woman,
* Patient carrying a pacemaker,
* Patients participating in another clinical study,
* Against indication to the realization of an MRI,
* Patient with a fistula with insufficient drainage, against indicating the removal of the stem (congestive fistula, oozing, with internal and / or external congestive orifices).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-04-17 (Actual); Primary Completion 2020-10-05 (Actual); Study Completion 2022-10-05 (Actual)

PRIMARY OUTCOMES:
Clinical healing of an anal fistula | 6 month
  Clinical healing of an anal fistula, 6 months after radiofrequency treatment: A fistula is clinically healed if there is no drain, the external and internal openings are non-inflammatory, clogged, and without flow.

SECONDARY OUTCOMES:
Clinical healing of an anal fistula, | 12 months
  Clinical healing of an anal fistula, 12 months after radiofrequency treatment: A fistula is clinically healed if there is no drain, the external and internal openings are non-inflammatory, clogged, and without flow.
evaluate anal continuation | 12 months
  evaluate anal continuation with SELF-EVALUATION QUESTIONNAIRE
Assessment of Feasibility of anal fistula treatment by radiofrequency | day 0 at inclusion
  Assessment of feasibility by measurement of anal fistula drying
Determination of the optimal settings | 12 months
  Evaluate the parameters of the probe (25 watts, 120 ° C, power 150 joules / 0,5 cm)
Patient satisfaction | 6 months
  self-assessment questionnaire with numerical scales
Patient satisfaction | 12 months
  self-assessment questionnaire with numerical scales
the rate and nature of post-operative complications | 12 months
  Number of Participants With Abnormal Values in MRI and Adverse Events That Are Related to Treatment
Evolution in MRI | 12 month
  If the MRI has eliminated an undrained pathway, a diverticulum greater than 10 mm, a hyper-intensity in T2 and after injection of Gadolinium.
Prognostic factors | 12 month
  Evaluate the prognostic factors of good or bad response to this treatment: type of fistula, settings of the probe and the drying of the fistula

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Abramowitz, MD, Principal Investigator — Clinique Blomet
Locations (4):
- France (4):
  - Chu Nantes, Nantes
  - Clinique Blomet, Paris
  - CHU Pontchaillou, Rennes
  - Hopital Bagatelle, Talence

IPD SHARING:
Plan to Share IPD: No